CLINICAL TRIAL: NCT01489813
Title: Phase II Randomized Placebo-Controlled Clinical Trial of Genistein in Reducing the Toxicity and Improving the Efficacy of Intravesical Therapy
Brief Title: Study of Genistein in Reducing Side Effects of Superficial Bladder Cancer Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Omer Kucuk, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00050273; EU2010-11 (Other: Winship Cancer Institute of Emory University); P30CA138292 (NIH)
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Results first posted 2024-07-25 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Genistein; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sugar pill (Placebo Comparator): Patients will be given placebo pills for 10 weeks.
  Interventions: Drug: Sugar pill
- Genistein supplement (Experimental): 30 mg of genistein supplement by mouth three times daily (PO TID) for 10 weeks.
  Interventions: Drug: Genistein

INTERVENTIONS:
Drug: Genistein — 30 mg of genistein supplement by mouth three times daily (PO TID).
  Other Names: Bonistein; I-Cool®
  Arms: Genistein supplement
Drug: Sugar pill — Sugar pills will be taken by mouth three times daily (PO TID).
  Other Names: Placebo pills
  Arms: Sugar pill

SUMMARY:
Patients with non-invasive bladder cancer are often treated with intravesical therapy in order to prevent the recurrence of bladder cancer. Intravesical therapy can cause many lower urinary tract symptoms, which can limit the dose of therapy and therefore efficacy of treatment. There have been a number of studies that suggest a chemical found in soy beans may be able to help with these side effects. This chemical is called genistein and can be extracted and given to study subjects in pill form. In this study, the investigators would like to have patients placed into two different groups. One group would take genistein and the other group would take a placebo, a sugar pill that looks like the genistein pill. In doing this study the investigators hope to explore the findings from other studies to see if lower urinary tract symptoms are reduced and to see if recurrence rates for patients are affected by genistein. The study would take about four and a half months total.

DETAILED DESCRIPTION:
Patients who are treated with bacillus Calmette-Guerin (BCG) intravesical therapy for non-muscle invasive (TaT1) Tis superficial bladder cancer often develop adverse effects (urinary tract symptoms) which limit the dose (and therefore the efficacy) of therapy and result in poor quality of life. Genistein is a nutritional supplement with anti-inflammatory properties which might help alleviate adverse effects of intravesical therapy that are due to inflammation. Additionally, genistein also has anti-tumor and immunopotentiating properties and has been shown to have no known side effects. Our hypothesis is that genistein given together with BCG intravesical therapy will reduce its adverse effects and improve the efficacy of therapy. Patients (N=88) scheduled for intravesical therapy will be randomly assigned to take 30 mg tablets PO TID of genistein supplement (N=44) or placebo (N=44) during therapy and one month post therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female gender
2. 18 years or older
3. Diagnosis of superficial bladder cancer
4. Scheduled for induction BCG intravesical therapy
5. Willing and able to give blood sample
6. Willing and able to fill out a pill diary to ensure compliance
7. Willing and able to sign informed consent
8. Birth control is not required for this study!

Exclusion Criteria:

1. Patients who are pregnant
2. Diagnosis of muscle-invasive bladder cancer
3. Unwillingness to follow study protocol and compliance procedures
4. HIV positive or immunocompromised
5. Receiving concurrent immunotherapy or chemotherapy
6. Presence of concurrent second cancer (active, not history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Department of Urology, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | Genistein Supplement
Started | 16 | 20
Completed | 13 | 17
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Genistein Supplement | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.3) | 71.2 (8.7) | 71.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 20 | 36
Number of Participants with Insurance [Count of Participants; unit: Participants] | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Urinary Symptoms as Determined by the The International Prostate Symptom Score (IPSS) Questionnaire Score.
Description: The change in severity of urinary symptoms as determined by the International Prostate Symptom Score (IPSS) questionnaire score. IPSS scores at 6 weeks of treatment will be compared to scores at baseline of treatment. Lower values indicate a better outcome.
  0 to 7 points: Mild symptoms 8 to 19 points: Moderate symptoms 20 to 35 points: Severe symptoms
Time Frame: At baseline and after 6 weeks of treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Sugar Pill | Genistein Supplement
Number analyzed (Participants) | 13 | 17
score on a scale | -2 [-3 to 2] | -3 [-4 to 2]

2. Secondary Outcome: Number of Participants With Cancer Recurrence Determined at 10-week Biopsy.
Description: A secondary study endpoint will be the presence of cancer and the rate of recurrence as determined by the 10-week biopsy or subsequent standard follow-up visits.
Time Frame: At 10 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Genistein Supplement
Number analyzed (Participants) | 14 | 18
Participants | 7 | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sugar Pill | Genistein Supplement
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 3/16 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=16) | Genistein Supplement (N=20)
Hospitalization (Infections and infestations) | 3 (3) | 3 (3)
UTI (Renal and urinary disorders) | 1 (1) | 1 (1)
Kidney infection (Renal and urinary disorders) | 0 (0) | 1 (1)
infection after urological surgical procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
coronovirus (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Actual enrollment was 36 subjects as reflected in the study data. Accrual did not meet the projected enrollment number due to lack of interest amongst patients and insufficient population within clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT01489813/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT01489813/ICF_000.pdf